CLINICAL TRIAL: NCT06938789
Title: The Impact of Bleeding on Delirium Outcomes in Older Patients With Hip Fractures: A Single-Blind, Randomized Controlled Trial - The IMPROVE-HIP Study
Brief Title: How Bleeding Affects Delirium in Older Patients With Hip Fractures: The IMPROVE-HIP Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Gødstrup Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JKB-1-2025
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Bleeding; Hip Fracture; Delirium - Postoperative
Keywords: Hip fracture; Delirium; Blood transfusion
MeSH Terms: conditions — Hemorrhage; Hip Fractures; Emergence Delirium; Delirium | interventions — Blood Transfusion; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Vital parameters, delirium screening, and blood samples are collected three times a day. If the hemoglobin level falls below our threshold, a blood transfusion is administered without delay.
  Interventions: Other: Blood Transfusion
- Control group (Placebo Comparator): The patients recieve standard care. To maintain patient blinding vital parameters, delirium screening, and blood samples are collected three times a day, just as in the intervention group, but their analysis is delayed to avoid influencing treatment decisions.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Blood Transfusion — Blood transfusion is given without delay (within 4 hours) in case of hemoglobin below our threshold.
  Arms: Intervention group
Other: Standard care — These patients recieve our standard care including blood transfusion as usual. Vital parameters and delirium screening are collected three times a day.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate whether early detection of bleeding and prompt blood transfusions can help prevent delirium in patients aged 75 and older who are admitted to the hospital with hip fractures. The main question the trial aims to answer is:

• Do patients aged 75 and older with hip fractures benefit from quicker treatment of anaemia (low blood count) to reduce the risk of delirium?

Researchers will compare early diagnosis and treatment of bleeding with standard care to determine if it helps lower the risk of developing delirium.

Participants will:

* Undergo blood tests and have their vital signs checked, as well as be screened for delirium three times a day for the first 48 hours after surgery.
* Receive blood transfusions promptly if their haemoglobin levels drop below a specified threshold.
* Have a follow-up visit at 30 days to assess their memory and overall quality of life.
* Have another follow-up at 90 days to check for hospital readmissions and survival

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture

Exclusion Criteria:

* Pathological hip fracture
* Periprosthtic fracture
* Unable to speak or understand Danish
* Does not wish to recieve blood transfusion
* If the investigator finds the patient unable to cooperate to the study (e.g. in case of severe dementia and externalizing behaviour)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Delirium | From enrollment to 48 hours after surgery
  Occurence of delirium will be evaluted using screening methods three times a day.

SECONDARY OUTCOMES:
Change from baseline in Quality of Life | Will be evaluated at the 30 day follow-up
  The overall Quality of life will be assed by the Overall Quality of life Depression List (OQoL-DL). It will be used to asses patients in both groups at the 30 day follow-up.
Cognitive status | Will be evaluated at the 30 day follow-up.
  Short Portable Mental Status Questionnaire (SPMSQ). Sum score 0-10, higher scores indicates cognitive impariment. The SPMSQ will be used to assess cognitve status in patients in both groups at follow-up.
Readmission rate | Within 90 days after surgery
  Readmission within 90 days after surgery. Readmission is defined as any uplanned, acute rehospitalisation in this period.
90-day mortality | 90 days after surgery.
  Mortality within the first 90-days after surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Gødstrup Hospital, Department of internal medicine, Herning, Central Jutland

IPD SHARING:
Plan to Share IPD: No